CLINICAL TRIAL: NCT03607214
Title: Longterm Effects of Expectations on Mood: An Experimental Investigation
Brief Title: Longterm Effects of Expectations on Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-15k
Record Dates: First submitted 2018-06-16; First posted 2018-07-31 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Expectations Group (Experimental): Participants receive a nasal spray that is in fact a placebo. However, they are told that it protects from experiencing negative emotions and generally improves their mood. They take the nasal spay in the laboratory and on seven consecutive days. Participants watch two film sequences that are supposed to induce sadness.
  Interventions: Other: Placebo
- No-treatment control group (No Intervention): Participants do not receive the nasal spray. Participants watch two film sequences that are supposed to induce sadness.

INTERVENTIONS:
Other: Placebo — Placebo nasal spray
  Film Sequence
  Arms: Positive Expectations Group

SUMMARY:
The study tries to identify whether positive expectations, induced with a placebo nasal-spray, have short- and longterm effects on participant's mood.

DETAILED DESCRIPTION:
Healthy volunteers are informed that a new application method for a well-known antidepressant would be tested. They will randomly be assigned to the experimental group (taking the antidepressant which is in fact an active placebo) or the control group (not taking a placebo). Then participants watch a well established film sequence to induce sadness. Sadness is assessed before and after receiving the nasal spray and watching the film sequence. In the seven consecutive days the participant's mood is assessed each day, only the experimental group is taking the placebo each day. Afterwards participants will watch another sad film sequence and sadness will be assessed before and afterwards.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* fluent in German language

Exclusion Criteria:

* mental disorders
* allergic to capsaicin
* allergic to sesame oil
* intake of psychopharmacological drugs
* intake of illegal drugs in the last two weeks
* consumption of alcohol in the last twelve hours
* students in medicine, pharmacy, or psychology
* completed studies in medicine, pharmacy or psychology

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS-X) | Directly before and after watching the film sequence and on the following seven days, each assessment is taking four minutes, in total 36 minutes.
  Items of PANAS-X: Sadness Score ("sad", "blue", "downhearted", "alone", "lonely") and Items "Surprised", "concentrating", "happy". All Items will be rated on a visual analogue scale from 0 (not at all) to 10 (very much).

SECONDARY OUTCOMES:
Coping with stress and daily hassles, general mood and concentration. | On seven consecutive days, each assesment is taking 3-5 minutes, in total 21 to 35 minutes
  The following Items are developed by the authors and will also be rated on a visual analogue scale (VAS) from 0 to 10.
  "How do you feel at the moment"? "How did you feel yesterday?" "How stress-resistent did you feel yesterday?" "How stress-resistant do you feel at the moment?"

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps-Univeristy of Marburg
Locations (1):
- Philipps-Universität Marburg, Marburg, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No